CLINICAL TRIAL: NCT04568291
Title: Clinical Reasearch on Three Dimensional Bionic Capture Network Circulating Tumor Cell in Lung Caner Patients With Bone Metastases
Brief Title: CTC in Lung Caner Patients With Bone Metastases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Zhao Hui, Clinical Professor, Shanghai 6th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTC01
Record Dates: First submitted 2020-03-06; First posted 2020-09-29 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Lung Cancer; Bone Metastases; Single Cell Sequencing Technology
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- routine treatment (Active Comparator): routine treatment
  Interventions: Other: routine treatment
- model treatment (Experimental): model treatment
  Interventions: Other: model treatment

INTERVENTIONS:
Other: model treatment — the treatment decisions were decided by Machine Learning （ML） model in model treatment group
  Arms: model treatment
Other: routine treatment — the treatment decisions were decided by multi-disciplinary team （MDT）
  Arms: routine treatment

SUMMARY:
1. Evaluate the feasibility of single cell sequencing technology based on three-dimensional bionic capture network;
2. To build a risk prediction model of bone related events based on single cell sequencing;
3. To verify the risk prediction model of bone related events by single cell sequencing;
4. To verify the comprehensive treatment of non-small cell lung cancer ( NSCLC) bone metastases.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-75 years
2. pathology-proven diagnosis of lung cancer and radiographical/pathological evidence of BM
3. no previous treatment for BM
4. good general condition (Eastern Cooperative Oncology Group, ECOG Performance scores: 0-2) with an estimated survival time > 3 months.

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
SREs（Skeletal related events） | 1 year
  occurance of SREs，including bone pain, pathological fractures, spinal cord compression, hypercalcemia, and the need for surgery or radiotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Sixth People'S Hospital, Shanghai, Other (Non U.s.), China